CLINICAL TRIAL: NCT00993915
Title: Non Interventional (NI) Open Label Prospective Study On Liprimar (Atorvastatin) In Patients With Coronary Heart Disease (CHD) And High Risk Of Cardiovascular Complications
Brief Title: Study On Liprimar (Atorvastatin) In Patients With Coronary Heart Disease (CHD) And High Risk Of Cardiovascular Complications
Acronym: LIGHT
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A2581185
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Results first posted 2012-12-20 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Cardiovascular Diseases; Coronary Artery Disease
Keywords: Coronary Artery Disease; Hyperlipidemia; Atorvastatin
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Hyperlipidemias | interventions — Atorvastatin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Main group: Newly diagnosed or known coronary artery disease and known dislipidemia and high risk of cardiovascular complications
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin, 10- 80 mg, once daily, 6 month treatment

SUMMARY:
In which CHD patients with high risk of CV complications are different doses of LIPRIMAR used? For this purpose, data on hyperlipidemia will be elicited over and above the basic nosographic and demographic data, concomitant diseases and cardiovascular risk factor.

ELIGIBILITY:
Inclusion Criteria:

* Patients, who eligible to sign informed consent;
* Patients with indications to lipid lowing therapy, according to local product document.
* Patients with CHD and high risk of CV complications (Diabetes Mellitus II, Myocardial Infarction, Heart Failure, Arterial Hypertension, ets) will be included into study;
* Patients with LDL levels: > 3,5 mmol/l

Exclusion Criteria:

* Individual intolerance of atorvastatin, in accordance to local product document.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Coronary atery disease, prevention of high risk cardiovascular complications with statins.
Sampling Method: Non-Probability Sample
Enrollment: 687 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581185&StudyName=Study%20On%20Liprimar%20%28Atorvastatin%29%20In%20Patients%20With%20Coronary%20Heart%20Disease%20%28CHD%29%20And%20High%20Risk%20Of%20Cardiovascular%20Complications

RESULTS

PARTICIPANT FLOW:
Groups:
- Atorvastatin: The use and dosage recommendations for Atorvastatin (Liprimar) were in accordance with the Local Product Development document. The recommended starting dose was 10 milligrams (mg) once daily, dosages adjusted as needed at intervals of 4 weeks or more, with a maximum dosage of 80 mg once daily.
Period: Overall Study
Arm/Group | Atorvastatin
Started | 687
Completed | 678
Not Completed | 9
Not completed — Insufficient clinical response | 3
Not completed — Withdrawal by Subject | 2
Not completed — Other | 1
Not completed — Ongoing | 3

BASELINE CHARACTERISTICS:
Arm/Group | Atorvastatin
Number analyzed (Participants) | 687
Age, Customized [Number; unit: participants]
  Between 18 and 44 years | 35
  Between 45 and 64 years | 493
  Greater than or equal to (≥) 65 years | 159
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 283
  Male | 404
Total cholesterol [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] — Number of participants with available data = 673
  milligrams per deciliter (mg/dL) | 271.69 (61.99)
Low-density lipoprotein (LDL) cholesterol [Mean (Standard Deviation); unit: mg/dL] — Number of participants with available data = 661
  mg/dL | 179.09 (54.19)
High-density lipoprotein (HDL) cholesterol [Mean (Standard Deviation); unit: mg/dL] — Number of participants with available data = 633
  mg/dL | 48.37 (20.14)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] — Number of participants with available data = 664
  mg/dL | 207.56 (145.61)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving LDL Level Less Than or Equal to (≤) 100 mg/dL at the 6 Month Visit
Time Frame: Month 6
Population: Full analysis set (FAS) population: all participants who received at least one dose of Atorvastatin (Liprimar) during the observation period and who had at least 1 post-baseline efficacy evaluation. Number of participants analyzed (N)= participants with evaluable data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atorvastatin
Number analyzed (Participants) | 592
percentage of participants | 51.52 [47.50 to 55.52]

2. Secondary Outcome: Percentage of Participants Achieving LDL Level ≤ 100 mg/dL at the 1 Month Visit
Time Frame: Month 1
Population: Not analyzed; LDL data not collected at 1 Month visit, time point erroneously identified for this outcome measure.
Arm/Group | Atorvastatin
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline in Lipid Parameters
Description: Lipid parameters include HDL cholesterol, LDL cholesterol, total cholesterol, and total triglycerides. Change = Month 6 value minus baseline
Time Frame: Month 6
Population: FAS Population. Number of participants analyzed (N) = participants with evaluable data; n = number of participants with evaluable data for the specific category. Change at Month 3 not analyzed; Month 3 visit not part of final protocol, time point erroneously identified for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Atorvastatin
Number analyzed (Participants) | 593
mg/dL
  Change at Month 6 in Total cholesterol, n=593 | -98.06 [-102.58 to -93.53]
  Change at Month 6 in LDL, n=583 | -76.84 [-80.49 to -73.19]
  Change at Month 6 in HDL, n=562 | 3.15 [1.61 to 4.70]
  Change at Month 6 in Triglycerides, n=585 | -70.57 [-80.73 to -60.41]

4. Secondary Outcome: Percent Change From Baseline in Lipid Parameters
Description: Percent change from baseline calculated as: 100*(change at Month X)/(baseline value).
Time Frame: Month 6
Population: FAS population. Number of participants analyzed (N) = participants with evaluable data; n = number of participants with evaluable data for the specific category. Percent change at Month 3 not analyzed; Month 3 visit not part of final protocol, time point erroneously identified for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Atorvastatin
Number analyzed (Participants) | 593
percent change
  Change at Month 6 in Total cholesterol, n=593 | -33.57 [-36.11 to -31.03]
  Change at Month 6 in LDL, n=583 | -40.66 [-42.15 to -39.17]
  Change at Month 6 in HDL, n=562 | 14.49 [11.38 to 17.60]
  Change at Month 6 in Triglyceride, n=585 | -23.05 [-25.58 to -20.51]

5. Other Pre Specified Outcome: Change From Baseline in Lipid Parameters at 1 Month
Description: as for outcome 3
Time Frame: Month 1
Population: Not analyzed; LDL data not collected at 1 Month visit, time point erroneously identified in registration for this outcome measure.
Arm/Group | Atorvastatin
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Percent Change From Baseline in Lipid Parameters at 1 Month
Description: Percent change from baseline calculated as: 100*(change at Month X)/(baseline value).
Time Frame: Month 1
Population: as for outcome 5
Arm/Group | Atorvastatin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Atorvastatin
Serious Adverse Events (participants affected / at risk) | 0/687
Other Adverse Events (participants affected / at risk) | 9/687
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin (N=687)
Abdominal pain (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Herpes zoster (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Cerebrovascular disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The end of study final status of 3 participants was not completed and therefore defaulted to ongoing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.